CLINICAL TRIAL: NCT01938898
Title: The NICOLA Recruitment Trial (NICOLA-RT): the Effect of Invitation Letters on Overall Recruitment in a Longitudinal Cohort Study in People Over Age of 50.
Brief Title: The NICOLA Recruitment Trial (NICOLA-RT)
Acronym: NICOLA-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Lisa Maguire, Research Fellow, Queen's University, Belfast
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 12/23
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy Cohort
Keywords: Randomized trial; Invitation letter; Recruitment; Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Potential NICOLA Participants (Other): All potential participants identified through the sampling strategy and contacted to take part in the NICOLA study
  Interventions: Other: Invitation letter randomisation

INTERVENTIONS:
Other: Invitation letter randomisation — There are 12 versions of the invitation letter. Three aspects of the letter will be adapted: (1) Gender of the signatory i.e. male, female or gender neutral (signed from the NICOLA team) (2) Description of NICOLA as a 'study' or 'project' and (3) Inserting a sentence guaranteeing the participants confidentially or not having this in the letter (but will still appear in the Patient Information Sheet). The twelve versions are as follows:
  1. Male & Study & Confidentiality
  2. Male & Study
  3. Male & Project & Confidentiality
  4. Male & Project
  5. Female & Project & Confidentiality
  6. Female & Project
  7. Female & Study & Confidentiality
  8. Female & Study
  9. Neutral & Study & Confidentiality
  10. Neutral & Study
  11. Neutral & Project & Confidentiality
  12. Neutral & Project

SUMMARY:
The Northern Ireland Cohort for the Longitudinal Study of Ageing (NICOLA) is an opportunity to conduct methodology research relevant to many features of a large prospective study. NICOLA will begin in earnest in Northern Ireland in 2013 and is being conducted by a multidisciplinary team in the Centre for Public Health at Queen's University Belfast. It is an omnibus programme of research on ageing that will continue for at least 10 years and will recruit 8500 middle-aged people in Northern Ireland and follow them into old age, providing a comprehensive assessment of their physical and mental health, their lifestyles, and their social and economic decision making. NICOLA will look at how they perceive disability and health, and how this differs between well-off and disadvantaged groups. NICOLA will also study various genetic, biological and psychological factors, including how participants perceive risk and value their time, and the effect of this on their retirement behaviour (including how they manage their money and their health). People over the age of 50 will be invited to take part and asked to complete detailed interviews and questionnaires every 2 years and health assessments every 4 years.

The overall aim of this research is to examine the impact of differing invitation letters offered to participants on study recruitment rates.

DETAILED DESCRIPTION:
Recruiting, retaining and gathering complete data on participants in research projects, be they patients or health professionals, can be extremely difficult. These problems increase the risk that research will be abandoned before its true value is appreciated, or lead to delays in resolving uncertainty for decision makers, while further studies are done. Poor recruitment, retention and outcome collection frequently lead to many prospective studies being extended, increasing costs. Researchers need to use strategies that are themselves evidence-based. This study links with an existing longitudinal ageing study called NICOLA to provide evidence on what research participants prefer in relation to providing personal information through a self-completed questionnaire. NICOLA is a large study of people over the age of 50 that is being conducted in Northern Ireland. NICOLA is aiming to recruit 8500 people and will ask them questions about participation in social activities, including organised structured and informal activities; relationship quality; loneliness; stress; resilience; quality of life; alcohol intake; food poverty and assess their health and wellbeing. Participants in NICOLA agree to having an interviewer visit them at home to ask questions about their lives, complete questionnaires in their own time and attend a health assessment appointment. They also agree to being followed up over a course of at least 10 years.

The research described here will examine the impact of differing invitation letters offered to participants on study recruitment rates, with the following specific objectives:

* Understanding if the gender of the person signing the invitation letter has an effect on recruitment
* Exploring the potential impact of the use of describing the research as a 'study' or as a 'project'
* Understanding if discussing and guaranteeing confidentiality for the participants in the invitation letter has an impact on recruitment.

We will do this by randomly allocating each of the 13000 participants contacted by NICOLA to receive invitation letter by one of the following three choices using a 3x2x2 factorial design:

1. Gender of the signatory (male versus female versus neutral team signature)
2. Description of NICOLA (study versus project)
3. Guarantee of confidentiality (inserted versus removed)

We will then analyse the numbers of participants agreeing to join NICOLA and use this to determine which invitation letter is the most acceptable to the participants. This research will occur within the first 18 months of NICOLA, when all participants are being recruited.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 50 or over.
* Participants must be living in an non-institutionalised environment.
* Participants must be capable of providing informed consent.

Exclusion Criteria:

* Participants who are 49 or younger.
* Participants who are institutionalised.
* Participants who are not capable of providing informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Influence of invitation letter on participation rates. | Average two weeks
  Difference in participation rates in those receiving letters (1) through to (12)

SECONDARY OUTCOMES:
Influence of invitation letter on study retention | Average twelve months
  Assessing the retention in the first year of the study including: completion of interview; return of self-completion questionnaire and participation in the health assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Clarke, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Lisa Maguire, Belfast, Northern Ireland, United Kingdom